CLINICAL TRIAL: NCT01704066
Title: Interobserver Variation in Applying a Radiographic Definition for ARDS: Impact of a Training Set of Berlin ARDS Definition
Brief Title: Interobserver Variation in Applying a Radiographic Definition for Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: Society of Critical Care Medicine, China (Other)
Responsible Party: Principal Investigator, Bin Du, Professor and Director, Medical ICU, Peking Union Medical College Hospital
Other Study IDs: CCCCTG-2012-ARDS-01; 2012BAI11B05 (Other Grant/Funding Number: National Key Technology R&D Program Project 2012BAI11B05)
Record Dates: First submitted 2012-10-06; First posted 2012-10-11 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Chest radiograph; Berlin Definition; Inter-observer agreement
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Training and education

SUMMARY:
The original American-European Consensus Conference (AECC) definition of Acute Respiratory Distress Syndrome (ARDS) required bilateral infiltrates consistent with pulmonary edema on frontal chest X-ray (CXR), but there is poor inter-observer reliability in interpreting CXR using this definition among intensivists and radiologists.

As a result, the newly published Berlin definition of ARDS specified that the CXR criterion should include bilateral opacities consistent with pulmonary edema not fully explained by effusions, lobar/lung collapse, or nodules/masses on CXR.

In order to improve inter-observer agreement, the panel have also developed a set of CXRs judged as consistent, inconsistent, or equivocal for the diagnosis of ARDS.

The objective of this study is to investigate the impact of this training set on inter-observer reliability in applying the radiographic definition for ARDS.

DETAILED DESCRIPTION:
The study is composed of 3 phases:

Phase 1: All participants will be required to independently interpret a set of 12 CXRs, as provided by the consensus panel. The possible radiographic interpretations include consistent, inconsistent, or equivocal for the diagnosis of ARDS.

Phase 2: Training materials adapted according to the recently published Berlin definition of ARDS, with its expanded rationale and interpretation of all 12 CXRs, will be sent to all participants.

Phase 3: The same set of 12 CXRs, in different order, will be sent to all participants for interpretation for the second time.

ELIGIBILITY:
Inclusion Criteria:

* intensivists working in the participating ICUs

Exclusion Criteria:

* those who could not participate both questionnaire surveys
* those who have read the reference with the training set of CXRs before the study
* those who have already known the objective of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Intensivists working in the participating ICUs
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
inter-observer agreement in the interpretation of CXRs for the diagnosis of ARDS | immediately after reading the CXRs

SECONDARY OUTCOMES:
Impact of the training set on the inter-observer agreement on the interpretation of CXRs | difference of inter-observer agreement before and after the training course

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Peng JM, Qian CY, Yu XY, Zhao MY, Li SS, Ma XC, Kang Y, Zhou FC, He ZY, Qin TH, Yin YJ, Jiang L, Hu ZJ, Sun RH, Lin JD, Li T, Wu DW, An YZ, Ai YH, Zhou LH, Cao XY, Zhang XJ, Sun RQ, Chen EZ, Du B; China Critical Care Clinical Trial Group (CCCCTG). Does training improve diagnostic accuracy and inter-rater agreement in applying the Berlin radiographic definition of acute respiratory distress syndrome? A multicenter prospective study. Crit Care. 2017 Jan 20;21(1):12. doi: 10.1186/s13054-017-1606-4. PMID 28107822